CLINICAL TRIAL: NCT07191470
Title: Isoflurane Sedation Using AnaConDa® Device With Non-Invasive Ventilation for the Management of Acute Exacerbation of COPD
Brief Title: Safety and Efficacy of Inhaled Sedation in Management of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pandit Bhagwat Dayal Sharma, PGIMS, Rohtak (Other)
Responsible Party: Principal Investigator, Aman Ahuja, Dr Aman Ahuja, Assistant Professor, Department of Pulmonary and Critical care medicine, Pandit Bhagwat Dayal Sharma, PGIMS, Rohtak
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BREC/23/121
Record Dates: First submitted 2025-08-19; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: COPD; ANACONDA; ISOFLURANE; inhalational anesthesia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Isoflurane inhalation via Anaesthetic Conserving Device (AnaConDa)
  Interventions: Device: The Anaesthetic Conserving Device (AnaConDa)

INTERVENTIONS:
Device: The Anaesthetic Conserving Device (AnaConDa) — The Anaesthetic Conserving Device (AnaConDa) was developed to facilitate the use of volatile anesthetics like isoflurane and isoflurane in mechanically ventilated patients outside the operating room. The device functions as a passive vaporizer, conserving anesthetic agents and reducing environmental contamination. Studies have demonstrated that AnaConDa-based inhaled sedation offers several advantages over intravenous sedation like better hemodynamic stability, reduced systemic inflammation, and faster recovery times.

SUMMARY:
Brief Summary (Plain Language)

This study tests whether using a device called AnaConDa® to give a mild gas medicine (isoflurane) helps people with severe flare-ups of chronic obstructive pulmonary disease (COPD) breathe more easily without needing a breathing tube. People with COPD sometimes breathe too fast or not deeply enough during non-invasive ventilation (NIV), which can cause agitation and poor mask fit. We want to see if a light level of isoflurane sedation makes NIV more comfortable, reduces the chance of needing a breathing tube, and is safe to use.

Who Can Join Adults aged 18 years or older with a diagnosed COPD flare-up and "hypercapnic respiratory failure" (too much carbon dioxide in the blood) who need NIV are eligible.

People with severe liver problems, a history of a rare reaction to anesthesia (malignant hyperthermia), very low consciousness (Glasgow Coma Scale below 12), or certain facial injuries cannot join. Pregnant people and those who recently had airway surgery also cannot join.

What Happens During the Study If you agree, we will place a special mask connected to a ventilator and the AnaConDa® device to give isoflurane gas. The gas rate starts at 1.5 mL per hour and aims for a light sedation level where you are drowsy but easily awakened (RASS -1 to -2). We will monitor your heart rate, blood pressure, breathing rate, and oxygen levels every hour for 24 hours. We'll draw small blood samples at the start and again at 2, 6, 12, and 24 hours to check carbon dioxide and oxygen levels. You will be asked how comfortable you feel on a simple scale of 0 ("very uncomfortable") to 10 ("very comfortable") at each time point.

Possible Benefits and Risks You may feel more relaxed and better tolerate the breathing mask, which could help you avoid a breathing tube. Risks include too much sedation (making you hard to wake), low blood pressure, slow heart rate, or slowed breathing. If excessive sedation or any serious issue occurs, we will stop the isoflurane and provide immediate medical care. A safety team will review all serious events within 24 hours.

Voluntary Participation and Confidentiality Joining this study is your choice. You can stop at any time without affecting your standard medical care. All your data will be kept private and stored in a secure database. Results will be shared only in groups, so no one will know your identity.

If you have questions or want to join, please contact:

Dr. Dhruva Chaudhry Phone: +91-999-110-1616 Email: dhruvachaudhry@yahoo.co.in

DETAILED DESCRIPTION:
Detailed Description:

Acute exacerbations of chronic obstructive pulmonary disease (COPD) often lead to too much carbon dioxide in the blood and difficulty breathing. Non-invasive ventilation (NIV) can help avoid a breathing tube, but many patients become agitated or uncomfortable with the mask, limiting its success. Traditional sedatives may worsen breathing or build up in the body. Isoflurane is an inhaled anesthetic with bronchodilator properties that can be given in small, quickly adjustable doses using the AnaConDa® device in-line with an NIV circuit. This study will test whether light isoflurane sedation can safely improve NIV tolerance and reduce the need for intubation in COPD flare-ups.

The study investigators will enroll 20 adults (age ≥ 18) admitted with a confirmed COPD exacerbation and hypercapnic respiratory failure who meet medical criteria for BiPAP-mode NIV. After obtaining informed consent, each participant will receive isoflurane delivered at 1.5 mL/hour via a syringe pump connected to the AnaConDa® device placed between the ventilator's Y-piece and the patient's mask. The fresh gas flow will be set equal to each patient's minute ventilation plus 0.5 L/min. NIV settings will be adjusted for comfort and gas exchange: pressure support 8-20 cm H₂O (target 10 mL/kg ideal body weight), PEEP 4-6 cm H₂O, respiratory rate 12-16 breaths/min (I:E ratio 1:3-1:4), and FiO₂ 30-40% to maintain SpO₂ 88-94%.

Sedation will be titrated to a light level (Richmond Agitation Sedation Scale [RASS] -1 to -2). If a patient becomes overly sedated (RASS ≤ -3) or requires endotracheal intubation within 24 hours, this will be recorded as an intervention failure and isoflurane will be stopped immediately. Continuous monitoring will include pulse oximetry, electrocardiogram, and non-invasive blood pressure (every 15 minutes for the first hour, then hourly). Arterial blood gases will be drawn at baseline and at 2, 6, 12, and 24 hours. At each time point we will also record RASS score and ask the patient to rate comfort on a 0-10 visual analogue scale (VAS).

The primary outcome is the proportion of patients experiencing intervention failure (intubation or excessive sedation) within 24 hours. Secondary outcomes are changes over time in vital signs (heart rate, blood pressure, respiratory rate), arterial blood gas values (pH, PaCO₂, PaO₂), sedation depth (RASS), patient comfort (VAS), and safety events (hypotension, bradycardia, respiratory depression, serious adverse events). We will follow participants until hospital discharge or intubation.

An interim analysis after the first 10 patients will assess safety and futility. The trial will be halted early if more than 50% of participants meet failure criteria or if the serious adverse event rate exceeds 20%. Data will be analyzed on both an intent-to-treat and per-protocol basis. Continuous measures will be compared using paired t-tests or nonparametric equivalents; categorical outcomes will use Chi-square or Fisher's exact tests; time-to-intubation will be analyzed with Kaplan-Meier methods.

This study is approved by the Institutional Ethics Committee (BREC 23/121) and will follow ICH-GCP and Declaration of Helsinki guidelines. All participant data will be anonymized and stored in a secure electronic database. Participation is voluntary, and patients may withdraw at any time without affecting their standard medical care.

ELIGIBILITY:
Inclusion Criteria

1. A confirmed diagnosis of COPD who had been admitted to the ICU due to acute exacerbation and hypercapnic respiratory failure requiring non-invasive ventilation.

Exclusion Criteria:

1. Any known allergy or contraindication to isoflurane, including hypersensitivity to isoflurane or other volatile anaesthetics.
2. A history of malignant hyperthermia or hepatic dysfunction suspected to be linked to prior exposure to volatile anaesthetics.
3. contraindications for NIV were taken into account, such as severe respiratory failure necessitating immediate invasive mechanical ventilation, facial trauma, burns, or anatomical abnormalities preventing proper mask fit, uncontrolled vomiting or excessive airway secretions, pneumothorax, and neurological impairment with a Glasgow Coma Scale (GCS) score of less than 12 and difficulty in airway protection.
4. Patients with hemodynamic instability, including shock unresponsive to fluid resuscitation, severe arrhythmias, or refractory hypotension unmanageable with NIV alone.
5. Pregnant patients or individuals who had recently undergone upper airway surgery or tracheostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with intervention failure | From enrollment to the end of treatment at 7 days
  intervention failure (defined as endotracheal intubation or Richmond Agitation-Sedation Scale score ≤ -3)

SECONDARY OUTCOMES:
Change from baseline in heart rate | from enrollment to the end of intervention at 7days
  Absolute difference in heart rate (beats per minute) from the pre-intervention value.
Change from baseline in blood pressure | From enrollment to the end of intervention at 7 days
  Absolute difference in systolic arterial pressure (mmHg) and diastolic blood pressure from the pre-intervention value.
Change in respiratory rate after intervention | From enrollment to the end of intervention at 7 days
  Absolute difference in respiratory rate (breaths per minute) from the pre-intervention value.
Change in Richmond Agitation-Sedation Scale (RASS) score | From enrollment to the end of treatment at 7 days
  RASS score (range +4 to -5; lower scores indicate deeper levels of sedation).
Visual Analogue Scale for patient comfort | From enrollment to the end of intervention at 7 days
  Description: VAS score (0 to 10; higher scores indicate greater comfort during NIV).

CONTACTS AND LOCATIONS:
Locations (1):
- Pandit Bhagwat Dayal Sharma Postgraduate Institute of Medical Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT07191470/Prot_SAP_ICF_000.pdf